CLINICAL TRIAL: NCT06454617
Title: Comparative Evaluation of Phantomless Calibration Methods to Quantify Bone Mineral Density for Opportunistic Analysis of CT Scans
Brief Title: Calibr-Ì: Comparative Evaluation of Phantomless Calibration Methods to Quantify Bone Mineral Density for Opportunistic Analysis of CT Scans
Acronym: Calibr-Ì
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Auckland Hospital - Greenlane Clinical Centre - National Women's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Calibr-I
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Phantoms, Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients that require a TC scan.
  Interventions: Other: Phantom

INTERVENTIONS:
Other: Phantom — The patients will be simultaneously scanned with a QCT phantom

SUMMARY:
Osteoporosis is a systemic disease characterized by a reduction in bone mineral density (BMD) and qualitative alteration of the skeleton, resulting in increased bone fragility and fracture risk. The epidemiological impact of osteoporosis is extremely high. Proper diagnosis and clinical management of osteoporosis are critical to reducing the incidence of fragility fractures and preventing their complications. The diagnosis is generally confirmed by instrumental analysis of bone mineral density. The standard method is X-ray bone densitometry (DXA), which allows diagnosis based on criteria defined by the World Health Organization (WHO) by virtue of the T-score. DXA is a relatively quick and inexpensive examination with low exposure to ionizing radiation. However, this method has limitations in detecting fracture risk, and in addition, not all patients are properly referred for DXA services, which, among other things, require specific criteria to be reimbursed by the National Health System. Currently, computed tomography (CT) scanning is the most widely used three-dimensional diagnostic modality in clinical practice, and the number of investigations performed in high-income countries is continuously growing. Quantitative assessment of bone mineral density by CT is possible by proper calibration of the machine for the purpose of converting the CT numbers (or Hounsfield units) measured by the scanner into BMD units.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* All ethnicities.
* Age equal or above 18 years.
* Any clinical indication (no specific pathology is required) for a CT scan of the lumbosacral spine or abdomen in which the entire lumbar spine (L1 to L5), paravertebral muscles, abdominal aorta, and subcutaneous adipose tissue are visible.
* Ability to give informed consent.

Exclusion Criteria:

* General contraindications to CT examination, including pregnancy or body weight/size exceeding scanner limits.
* Severe degenerative manifestations of the lumbosacral spine.
* Severe scoliosis of the lumbosacral spine.
* Surgical hardware that prevents adequate CT scanning.
* Oncologic pathology in progress or in recent history.
* Any other situation deemed incompatible with the study by the designated physician or investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve a population of patients undergoing CT scans including the lumbar spine at the Diagnostic and Interventional Radiology Unit of each participating center. In CT scans requiring the administration of contrast medium, only the non-contrast-enhanced images will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of different internal calibration methods | At baseline (Day 0)
  Compare the different methods of internal or phantomless calibration described in the literature with synchronous and asynchronous calibration in a population of patients undergoing CT scans that include the lumbar spine to assess their feasibility.

SECONDARY OUTCOMES:
Definition of performance of internal calibration methods | At baseline (Day 0)
  Define the performance of various internal or phantomless calibration methods for the purpose of identifying the most appropriate and reliable technique.
Optimization of existing internal calibration methods | Through study completion, up to 2 years
  Optimize existing internal calibration methods, and eventually define a new phantomless targeted calibration protocol based on the results of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- The Rizzoli Orthopaedic Institute, Bologna, Bo, Italy
- Auckland Hospital - Greenlane Clinical Centre - National Women's Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rossini M, Adami S, Bertoldo F, Diacinti D, Gatti D, Giannini S, Giusti A, Malavolta N, Minisola S, Osella G, Pedrazzoni M, Sinigaglia L, Viapiana O, Isaia GC. Guidelines for the diagnosis, prevention and management of osteoporosis. Reumatismo. 2016 Jun 23;68(1):1-39. doi: 10.4081/reumatismo.2016.870. PMID 27339372
- [Result] Willers C, Norton N, Harvey NC, Jacobson T, Johansson H, Lorentzon M, McCloskey EV, Borgstrom F, Kanis JA; SCOPE review panel of the IOF. Osteoporosis in Europe: a compendium of country-specific reports. Arch Osteoporos. 2022 Jan 26;17(1):23. doi: 10.1007/s11657-021-00969-8. PMID 35079919
- [Result] Engelke K, Lang T, Khosla S, Qin L, Zysset P, Leslie WD, Shepherd JA, Shousboe JT. Clinical Use of Quantitative Computed Tomography-Based Advanced Techniques in the Management of Osteoporosis in Adults: the 2015 ISCD Official Positions-Part III. J Clin Densitom. 2015 Jul-Sep;18(3):393-407. doi: 10.1016/j.jocd.2015.06.010. PMID 26277853
- [Result] Michalski AS, Besler BA, Michalak GJ, Boyd SK. CT-based internal density calibration for opportunistic skeletal assessment using abdominal CT scans. Med Eng Phys. 2020 Apr;78:55-63. doi: 10.1016/j.medengphy.2020.01.009. Epub 2020 Feb 12. PMID 32059948